CLINICAL TRIAL: NCT01493947
Title: Efficacy and Safety of CD5024 1% Cream Versus Metronidazole 0.75% Cream in Subjects With Papulopustular Rosacea Over 16 Weeks Treatment, Followed by a 36-week Extension Period.
Brief Title: CD5024 1% [Ivermectin 1%] Cream Versus Metronidazole 0.75% Cream in Papulopustular Rosacea (PPR) Study
Acronym: ATTRACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.40173
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — Ivermectin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivermectin 1% cream (Experimental)
  Interventions: Drug: Ivermectin 1% cream
- Metronidazole 0.75% cream (Active Comparator)
  Interventions: Drug: Metronidazole 0.75% cream

INTERVENTIONS:
Drug: Ivermectin 1% cream — Ivermectin 1% cream applied once daily on the face during 16-week plus 36-week extension period.
  Other Names: Soolantra
  Arms: Ivermectin 1% cream
Drug: Metronidazole 0.75% cream — Metronidazole 0.75% cream applied twice daily on the face during 16-week plus 36-week extension period.
  Other Names: Metronidazole
  Arms: Metronidazole 0.75% cream

SUMMARY:
Study objectives:

* To compare efficacy and safety of Ivermectin 1% cream versus metronidazole 0.75% cream in subjects with papulopustular rosacea after 16-week topical treatment.
* And to compare, for subjects initially successfully treated by 16 weeks treatment, Ivermectin 1 % cream versus metronidazole 0.75% cream during a 36-week extension period by assessing, the time of first relapse, the relapse rate, and the number of days free of treatment

ELIGIBILITY:
Inclusion Criteria:

* Subjects with papulopustular rosacea scored 3 (moderate) or 4 (severe) according to the Investigator Global Assessment (IGA),
* Subjects with at least 15 but not more than 70 inflammatory lesions (papules and pustules) on the face.

Exclusion Criteria:

* Subjects with particular forms of rosacea (rosacea conglobate, rosacea fulminant, isolated rhinophyma, isolated pustulosis of the chin) or other facial dermatoses that may be confounded with papulopustular rosacea, such as peri oral dermatitis, facial keratosis pilar, or seborrheic dermatitis and acne,
* Subjects with rosacea with more than two nodules on the face.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 962 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- Bulgaria (3):
  - Galderma Investigational Site, Pleven
  - Galderma Investigational Site, Plovdiv
  - Galderma Investigational Site, Sofia
- Czechia (6):
  - Galderma Investigational Site, Chomutov
  - Galderma Investigational Site, Hradec Králové
  - Galderma Invetigational site, Olomouc
  - Galderma Investigational Site, Pardubice
  - Galderma Investigational Site, Prague
  - Galderma Investigational Site, Slaný
- France (5):
  - Galderma Investigational Site, Bordeaux
  - Galderma Investigational Site, Brest
  - Galderma Investigational Site, Cannes
  - Galderma Investigational Site, Nice
  - Galderma Investigational Site, Saint-Etienne
- Germany (13):
  - Galderma Investigational Site, Augsburg
  - Galderma Investigational Site, Berlin
  - Galderma Investigational Site, Bonn
  - Galderma Investigational Site, Darmstadt
  - Galderma Investigational Site, Dresden
  - Galderma Investigational Site, Hamburg
  - Galderma Investigational Site, Langenau
  - Galderma Investigational Site, Mahlow
  - Galderma Investigational Site, Mainz
  - Galderma Investigational Site, Munich
  - Galderma Investigational Site, Münster
  - Galderma Investigational Site, Tübingen
  - Galderma Investigational Site, Wuppertal
- Hungary (7):
  - Galderma Investigational Site, Budapest
  - Galderma Investigational Site, Debrecen
  - Galderma Investigational Site, Miskolc
  - Galderma Investigational Site, Pécel
  - Galderma Investigational Site, Szeged
  - Galderma Investigational Site, Szekszárd
  - Galderma Investigational Site, Szolnok
- Poland (5):
  - Galderma Investigational Site, Bialystok
  - Galderma Investigational Site, Gdansk
  - Galderma Investigational Site, Krakow
  - Galderma Investigational Site, Warsaw
  - Galderma Investigational Site, Wroclaw
- Romania (5):
  - Galderma Investigational Site, Brasov
  - Galderma Investigational Site, Bucharest
  - Galderma Investigational Site, Craiova
  - Galderma Investigational Site, Târgu Mureş
  - Galderma Investigational Site, Timișoara
- Russia (4):
  - Galderma Investigational Site, Chelyabinsk
  - Galderma Investigational Site, Lipetsk
  - Galderma Investigational Site, Moscow
  - Galderma Investigational Site, Nizhny Novgorod
- Ukraine (5):
  - Galderma Investigational Site, Dnipropetrovsk
  - Galderma Investigational Site, Donetsk
  - Galderma Investigational Site, Kiev
  - Galderma Investigational Site, Lviv
  - Galderma Investigational Site, Uzhhorod
- United Kingdom (4):
  - Galderma Investigational Site, Berkshire
  - Galderma Investigational Site, Bexhill-on-Sea
  - Galderma Investigational Site, London
  - Galderma Investigational Site, Nuneaton

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivermectin: Ivermectin applied once daily on the face during 16-week
- Metronidazole 0.75% Cream: Metronidazole 0.75% cream applied twice daily on the face during 16-week
Period: Period A Efficacy and Safety Data
Arm/Group | Ivermectin | Metronidazole 0.75% Cream
Started | 478 | 484
Completed | 446 | 456
Not Completed | 32 | 28
Period: Period B Extension Period
Arm/Group | Ivermectin | Metronidazole 0.75% Cream
Started | 399 (Only 399 /446 subjects were eligible to enter in Period B (i.e IGA=0 or1 at end of Period A).) | 358 (358 / 456 subjects were eligible to enter in Period B (i.e IGA =0 or 1 at end of Period A).)
Completed | 366 | 326
Not Completed | 33 | 32

BASELINE CHARACTERISTICS:
Groups:
- Ivermectin: Ivermectin: Ivermectin applied once daily on the face during 16-week plus 36-week extension period.
- Total: Total of all reporting groups
Arm/Group | Ivermectin | Metronidazole 0.75% Cream | Total
Number analyzed (Participants) | 478 | 484 | 962
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 394 | 398 | 792
  >=65 years | 84 | 86 | 170
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311 | 316 | 627
  Male | 167 | 168 | 335
Region of Enrollment [Number; unit: participants]
  Czech Republic | 40 | 40 | 80
  Russian Federation | 39 | 35 | 74
  Romania | 57 | 52 | 109
  Hungary | 76 | 84 | 160
  Ukraine | 30 | 30 | 60
  Poland | 57 | 57 | 114
  United Kingdom | 16 | 19 | 35
  Bulgaria | 20 | 17 | 37
  France | 31 | 36 | 67
  Germany | 112 | 114 | 226

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Inflammatory Lesions From Baseline to Week 16
Description: Efficacy of Ivermectin versus Metronidazole as determined by the percent change in inflammatory lesions after a 16-week treatment period
Time Frame: Baseline and Week 16
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ivermectin | Metronidazole 0.75% Cream
Number analyzed (Participants) | 478 | 484
percentage of change | -83 (26) | -73.7 (39.7)

2. Other Pre Specified Outcome: Time to Relapse
Description: Relapse define as time elapsed between Week 16 and first reoccurrence of Investigator Global assessement (IGA) at '2 (mild)' , '3 (moderate)' or '4 (severe)'.
Time Frame: Week 16 up to Week 52
Measure: Median (95% Confidence Interval); unit: Median days to relapse
Groups:
- CD5024: CD5024: CD5024 applied once daily on the face during 16-week plus 36-week extension period.
Arm/Group | CD5024 | Metronidazole 0.75% Cream
Number analyzed (Participants) | 399 | 358
Median days to relapse | 115 [113 to 165] | 85 [85 to 113]

ADVERSE EVENTS:
Description: One subject received Ivermectin in Period A,but after relapse received metronidazole in Period B. This subject was counted in each group, but the Adverse Events (AEs) are counted according to their onset date.
Groups:
- Ivermectin 1% Cream Period A: Ivermectin applied once daily on the face during 16-week
- Metronidazole 0.75% Cream Period A: Metronidazole 0.75% cream applied twice daily on the face during 16-week
- Ivermectin 1% Cream Period B: 36-week extension period :only subjects with an IGA of 0 or 1 at Week 16 (i.e., at the last visit of Period A) were eligible
- Metronidazole 0.75% Cream Period B: 36-week extension period : only subjects with an IGA of 0 or 1 at Week 16 (i.e., at the last visit of Period A) were eligible.
Arm/Group | Ivermectin 1% Cream Period A | Metronidazole 0.75% Cream Period A | Ivermectin 1% Cream Period B | Metronidazole 0.75% Cream Period B
Serious Adverse Events (participants affected / at risk) | 8/478 | 5/484 | 10/399 | 11/359
Other Adverse Events (participants affected / at risk) | 101/478 | 100/484 | 110/399 | 91/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin 1% Cream Period A (N=478) | Metronidazole 0.75% Cream Period A (N=484) | Ivermectin 1% Cream Period B (N=399) | Metronidazole 0.75% Cream Period B (N=359)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitello-Intestinal Duct Remnant (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular Degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema Infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain Herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoathritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolitiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Femoral Artery Occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Whiplash Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin 1% Cream Period A (N=478) | Metronidazole 0.75% Cream Period A (N=484) | Ivermectin 1% Cream Period B (N=399) | Metronidazole 0.75% Cream Period B (N=359)
Nasopharingitis (Infections and infestations) | 32 (32) | 29 (29) | 37 (37) | 39 (39)
Influenza (Infections and infestations) | 9 (9) | 10 (10) | 12 (12) | 6 (6)
Headache (Nervous system disorders) | 15 (15) | 11 (11) | 5 (5) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4) | 6 (6) | 5 (5)
Bronchitis (Infections and infestations) | 6 (6) | 4 (4) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 6 (6) | 4 (4) | 4 (4) | 7 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (6) | 4 (4) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 3 (3) | 5 (5) | 7 (7) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 4 (4) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 5 (5) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 5 (5) | 6 (6)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No